CLINICAL TRIAL: NCT06979531
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 in Adult Participants With Primary Sjogren's Disease With Moderate to Severe Systemic Disease Activity
Brief Title: Efficacy and Safety of IMVT-1402 in Adult Participants With Primary Sjogren's Disease With Moderate to Severe Systemic Disease Activity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMVT-1402-2801; 2025-520831-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Sjogren Disease; IMVT-1402

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Sponsor will also be blinded in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: IMVT-1402 Dose 1 (Experimental)
  Interventions: Drug: IMVT-1402
- Group 2: IMVT-1402 Dose 2 (Experimental)
  Interventions: Drug: IMVT-1402
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMVT-1402 — Administered once weekly by subcutaneous injection
  Arms: Group 1: IMVT-1402 Dose 1; Group 2: IMVT-1402 Dose 2
Drug: Placebo — Administered once weekly by subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a Phase 2b, multicenter, randomized, double-blinded, placebo-controlled study to assess the efficacy and safety of IMVT-1402 in adult participants with moderate to severe systemic primary Sjogren's disease (SjD).

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy, safety, and tolerability of IMVT-1402 compared to placebo, as measured by the change from baseline of Clinical European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (cliniESSDAI) at Week 24.

The total duration of study participation is expected to be up to 57 weeks for an individual participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of primary SjD for at least 12 months prior to the Screening Visit and meet classification criteria for primary SjS according to the 2016 American College of Rheumatology/ European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome at the time of screening.
* Participants with moderate to severe systemic disease activity as determined by a clinESSDAI total score ≥ 5 at the Screening Visit.
* Participants are seropositive for antibodies to Sjogren's Syndrome A (SSA)/Anti-Sjogren's Syndrome A (Ro) at the Screening Visit.
* Participants have residual salivary flow as measured by stimulated whole salivary flow rate ≥ 0.01 milliliters per minute (mL/min) at the Screening Visit.

Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Participants with a diagnosis of secondary SjD or an autoimmune disease other than primary SjD that constitutes the principal illness, including but not limited to, rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, dermatomyositis, pre-existing fibromyalgia or polymyositis, at the Screening Visit.
* Participants with a history of clinically significant monoclonal gammopathy, including but not limited to monoclonal gammopathy of undetermined significance, history of multiple myeloma or non-Hodgkin's lymphoma, or have an active malignancy or history of malignancy within 5 years prior to the Screening Visit.

Additional exclusion criteria are defined in the protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in clinESSDAI Score at Week 24 for IMVT-1402 Dose 1 compared to Placebo | Baseline and at Week 24
  The clinESSDAI is a tool used in clinical studies to measure the systemic disease activity in participants with primary Sjogren's syndrome.

SECONDARY OUTCOMES:
Proportion of clinESSDAI responders at Week 24 for IMVT-1402 Dose 1 compared to Placebo | Week 24
  A clinESSDAI responder is defined as participants having achieved clinESSDAI ≥ 4 points improvement from Baseline.
Change from Baseline in clinESSDAI score at Week 24 for IMVT-1402 Dose 2 compared to Placebo | Baseline, Week 24
Proportion of clinESSDAI responders at Week 24 for IMVT-1402 Dose 2 compared to Placebo | Week 24
  A clinESSDAI responder is defined as participants having achieved clinESSDAI ≥ 4 points improvement from Baseline.
Proportion of clinESSDAI responders at Week 48 for IMVT-1402 Dose 1 compared to Placebo | Week 48
  A clinESSDAI responder is defined as participants having achieved clinESSDAI ≥ 4 points improvement from Baseline.
Proportion of clinESSDAI responders at Week 48 for IMVT-1402 Dose 2 compared to Placebo | Week 48
  A clinESSDAI responder is defined as participants having achieved clinESSDAI ≥ 4 points improvement from Baseline.
Change from baseline in Physician General Assessment of Disease Activity (PhGA) score at Week 24 for IMVT-1402 Dose 1 compared to Placebo | Baseline and at Week 24
  The PhGA is a measure of the participant's current disease activity as assessed by the physician or another healthcare professional.
Change from baseline in PhGA score at Week 24 for IMVT-1402 Dose 2 compared to Placebo | Baseline and at Week 24
  The PhGA is a measure of the participant's current disease activity as assessed by the physician or another healthcare professional.

CONTACTS AND LOCATIONS:
Locations (121):
- United States (29):
  - Site Number - 1027, Covina, California
  - Site Number - 1007, El Cajon, California
  - Site Number - 1016, Menifee, California
  - Site Number - 1029, Thousand Oaks, California
  - Site Number - 1026, Upland, California
  - Site Number - 1014, Fort Collins, Colorado
  - Site Number - 1018, Hollywood, Florida
  - Site Number - 1021, Jupiter, Florida
  - Site Number - 1002, Miami, Florida
  - Site Number - 1004, Tamarac, Florida
  - Site Number - 1025, Tampa, Florida
  - Site Number - 1012, Chicago, Illinois
  - Site Number - 1033, Orland Park, Illinois
  - Site Number - 1030, Lake Charles, Louisiana
  - Site Number - 1028, New Orleans, Louisiana
  - Site Number - 1032, Canton, New York
  - Site Number - 1006, Mineola, New York
  - Site Number - 1013, Philadelphia, Pennsylvania
  - Site Number - 1015, Jackson, Tennessee
  - Site Number - 1000, Memphis, Tennessee
  - Site Number - 1001, Allen, Texas
  - Site Number - 1020, Amarillo, Texas
  - Site Number - 1022, Arlington, Texas
  - Site Number - 1019, Austin, Texas
  - Site Number - 1024, Grapevine, Texas
  - Site Number - 1011, Houston, Texas
  - Site Number - 1010, Houston, Texas
  - Site Number - 1023, Katy, Texas
  - Site Number - 1031, San Antonio, Texas
- Argentina (9):
  - Site number - 5005, Azcuénaga, Buenos Aires
  - Site Number - 5007, Capital Federal, Buenos Aires
  - Site Number - 5008, San Isidro, Buenos Aires
  - Site Number - 5004, San Miguel de Tucumán, Tucumán Province
  - Site Number - 5000, Buenos Aires
  - Site Number - 5002, Buenos Aires
  - Site Number - 5003, Buenos Aires
  - Site Number - 5001, Buenos Aires
  - Site number - 5006, Buenos Aires
- Brazil (6):
  - Site Number - 5506, Vitória, Espírito Santo
  - Site Number - 5504, Salvador, Estado de Bahia
  - Site Number - 5500, Juiz de Fora, Minas Gerais
  - Site Number - 5501, Curitiba, Paraná
  - Site Number - 5503, Porto Alegre, Rio Gtande Do Sul
  - Site Number - 5505, Porto Alegre, Rio Gtande Do Sul
- Canada (2):
  - Site Number - 2001, Sherbrooke, Quebec
  - Site Number - 2000, Trois-Rivières, Quebec
- Chile (8):
  - Site Number - 5706, Viña del Mar, Región de Valparaíso
  - Site Number - 5700, Santiago, Santiago de Chile
  - Site Number - 5702, Santiago, Santiago de Chile
  - Site Number - 5703, Santiago, Santiago de Chile
  - Site Number - 5701, Santiago, Santiago de Chile
  - Site Number - 5704, Santiago, Santiago de Chile
  - Site Number - 5705, Osorno
  - Site Number - 5707, Valdivia
- Colombia (5):
  - Site Number - 5800, Medellín, Antioquia
  - Site Number - 5804, Barranquilla, Atlántico
  - Site Number - 5803, Bogotá, Cundinamarca
  - Site Number - 5802, Chía, Cundinamarca
  - Site Number - 5801, Bucaramanga, Santander Department
- Germany (7):
  - Site Number - 6504, Bad Doberan
  - Site Number - 6506, Cologne
  - Site Number - 6500, Hamburg
  - Site Number - 6501, Hanover
  - Site Number - 6503, Heidelberg
  - Site number - 6502, Munich
  - Site Number - 6505, Munich
- Greece (2):
  - Site Number - 3901, Athens
  - Site Number - 3900, Athens
- Hungary (4):
  - Site Number - 7550, Budapest
  - Site Number - 7552, Hódmezővásárhely
  - Site Number - 7551, Kalocsa
  - Site Number - 7553, Székesfehérvár
- Italy (7):
  - Site Number - 6000, Catania
  - Site Number - 6001, Milan
  - Site Number - 6006, Naples
  - Site Number - 6002, Palermo
  - Site Number - 6005, Perugia
  - Site Number - 6003, Rome
  - Site Number - 6007, Salerno
- Mexico (8):
  - Site Number - 2602, Guadalajara, Jalisco
  - Site Number - 2604, Cuautitlán Izcalli, State of Mexico
  - Site Number - 2605, Toluca, State of Mexico
  - Site Number - 2607, Mérida, Yucatán
  - Site Number - 2601, Chihuahua City
  - Site Number - 2600, Mexico City
  - Site Number - 2606, Mexico City
  - Site Number - 2603, Mexico City
- Peru (4):
  - Site Number - 2400, Cayma, Arequipa
  - Site Number - 2401, Santiago de Surco, Lima region
  - Site Number - 2403, Lima
  - Site Number - 2402, Lima
- Poland (16):
  - Site Number - 3008, Bydgoszcz
  - Site Number - 3010, Krakow
  - Site Number - 3014, Lodz
  - Site Number - 3004, Lodz
  - Site Number - 3015, Lublin
  - Site Number - 3005, Lublin
  - Site Number - 3007, Poznan
  - Site Number - 3000, Poznan
  - Site Number - 3011, Siedlce
  - Site Number - 3006, Warsaw
  - Site Number - 3001, Warsaw
  - Site Number - 3003, Warsaw
  - Site Number - 3009, Warsaw
  - Site Number - 3012, Wołomin
  - Site Number - 3002, Wroclaw
  - Site Number - 3013, Wroclaw
- Romania (3):
  - Site Number - 7502, Brasov
  - Site Number - 7500, Bucharest
  - Site Number - 7501, Cluj-Napoca
- Spain (6):
  - Site Number - 7103, Bilbao
  - Site Number - 7106, Cadiz
  - Site Number - 7101, Córdoba
  - Site Number - 7102, Mérida
  - Site Number - 7100, Santa Cruz de Tenerife
  - Site Number - 7104, Valencia
- United Kingdom (5):
  - Site Number - 7004, Cambridge
  - Site Number - 7003, Liverpool
  - Site Number - 7002, London
  - Site Number - 7000, Swindon
  - Site Number - 7001, Truro

IPD SHARING:
Plan to Share IPD: No